CLINICAL TRIAL: NCT05519358
Title: Efficacy of Midsagittal Tongue Cross-section Area Measured by Ultrasound in Predicting Difficult Airway in Obesity Surgery Patients
Brief Title: Midsagittal Tongue Measurement to Predict Difficult Airways
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Suna Kara Gormus, Principal Investigator, Samsun University
Other Study IDs: SKara
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Difficult Airway; Ultrasonography
Keywords: Airway management; Ultrasonography; Tongue widht

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- difficult airway: difficult laryngoscopy; Cormack-Lehane grades 3 or 4 or Difficult intubation; Intubation Difficulty Scale (IDS)> 5 .IDS based on parameters known to be associated with difficult intubation
- non difficult airway: not difficult intubation or laryngoscopy

SUMMARY:
An unanticipated difﬁcult airway is a potentially life-threatening event during elective surgery or management of critical conditions. However, the common clinical screening tests, show low sensitivity and specificity with a limited predictive value. Recently, ultrasound has been used to identify difficult airway. Tongue volume is one of the parameters evaluated by ultrasound. In this study, we aim to evaluate the capacity of mid-sagittal tongue CSA and tongue width to predict difficult laryngoscopy and difficult intubation.

DETAILED DESCRIPTION:
Anatomical changes that adversely affect airway accessibility due to increased adipose tissue in obese patients make it difficult to establish an advanced airway by orotracheal intubation. Difficulty with airway management for anesthesia has potentially serious implications, as failure to secure a patent airway can result in hypoxic brain injury or death in a matter of minutes. There have been no effective methods to predict difficult airways accurately. Ultrasonography is a non-invasive, safe, and painless modality for evaluating soft tissues. In recent years, studies have been carried out on the parameters that can be used in determining the difficult airway with ultrasound. These include the distance from the skin to the epiglottis, the tongue thickness, the tongue volume, the mandibular condylar mobility, and the visibility of the hyoid. Few studies have whether midsagittal tongue cross section area and tongue width can also be used to predict difficult airways similarly to tongue volume. Therefore, this study was designed to evaluate the predictive value of accurately measured tongue thickness and cross-sectional tongue area using ultrasonography for predicting difficult tracheal intubation and difficult laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical condition I-II-III
* Patients are required general anesthesia with tracheal intubation for bariatric surgery.

Exclusion Criteria:

* Patients with maxillofacial deformity, trauma, or tumor
* Patients with identified difficult airway or difficult airway history
* Patients with cancellation of tracheal intubation for a non-difficult airway reason

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are18 to 90 years old and of either sex who required general anesthesia with tracheal intubation for bariatric surgery .
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
midsagittal tongue cross- sectional area | All of the enrolled patients received ultrasonic measurement in the operation room before anesthesia on the day of surgery.
  To evaluate the capability of midsagittal tongue cross- sectional area measured by ultrasound to predict difficult laryngoscopy and difficult intubation.
tongue width | All of the enrolled patients received ultrasonic measurement in the operation room before anesthesia on the day of surgery.
  To evaluate the capability of tongue widht measured by ultrasound to predict difficult laryngoscopy and difficult intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Suna KARAGÖRMÜŞ, Principal Investigator — Samsun Univercity
Locations (1):
- Samsun University Faculty of medicine, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moura ECR, Filho ASM, de Oliveira EJSG, Freire TT, da Cunha Leal P, de Sousa Gomes LMR, Servin ETN, de Oliveira CMB. Comparative Study of Clinical and Ultrasound Parameters for Defining a Difficult Airway in Patients with Obesity. Obes Surg. 2021 Sep;31(9):4118-4124. doi: 10.1007/s11695-021-05528-1. Epub 2021 Jul 5. PMID 34227021
- [Background] Alessandri F, Antenucci G, Piervincenzi E, Buonopane C, Bellucci R, Andreoli C, Alunni Fegatelli D, Ranieri MV, Bilotta F. Ultrasound as a new tool in the assessment of airway difficulties: An observational study. Eur J Anaesthesiol. 2019 Jul;36(7):509-515. doi: 10.1097/EJA.0000000000000989. PMID 31742568
- [Background] Yao W, Wang B. Can tongue thickness measured by ultrasonography predict difficult tracheal intubation? Br J Anaesth. 2017 Apr 1;118(4):601-609. doi: 10.1093/bja/aex051. PMID 28403413